CLINICAL TRIAL: NCT01186627
Title: Trial to Evaluate a Specified Type of Apgar (TEST-APGAR) Follow-Up Study
Brief Title: Trial to Evaluate a Specified Type of Apgar (TEST-APGAR) Follow Up Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Prof. Dr. Mario Ruediger, Dresden University of Technology, Department of Neonatology
Other Study IDs: Test-Apgar Follow-Up
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2010-10

CONDITIONS: Premature Birth; Mortality; Apgar Score
Keywords: Neurodevelopmental Impairment; Intraventricular hemorrhage; Retinopathy of prematurity; Mortality; Apgar Score
MeSH Terms: conditions — Premature Birth; Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A specified version of the Apgar-Score, that can be used in newborns under resuscitation, was developed and its value to predict chronic damage in preterm infants will be tested.

DETAILED DESCRIPTION:
Specifications of the individual items of the original Apgar score were suggested. These specifications slightly changed the Apgars' perspective, but did not alter the number of its components. The specified Apgar should therefore be easily applicable to every delivery room around the world. As a result of these specifications, the Apgar score will not express the efforts of the infant but describe its condition, independently of the requirements needed to achieve this condition. The advantage of the proposed definitions is the applicability in all infants, regardless of resuscitative efforts or gestational age.

To validate the accuracy of the specified version to predict neonatal mortality and long term neurological outcome in preterm infants the present prospective, observational study is planned. The study will test the hypothesis that the specified APGAR-score predicts mortality and morbidity better at 2 years of age than the conventional Apgar-score. Furthermore, the predictive reliability of the specified Apgar can be improved in combination with perinatal data respectively with the expanded Apgar version of the AAP/ACOG.

The primary outcome "condition at 2 years of age" is composed of death and a major neurological deficit. In this case "neurological deficit" is defined by the presence of one of the followings characteristics: index of mental development (Bayley Scale II) <85, blindness, deafness, cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* All preterm infants included in the TEST-APGAR Study

Exclusion Criteria:

* Missing parental Consent

Ages: 2 Years to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Former preterm infants with a gestational age below 32 weeks which have been included in the TEST-APGAR Study are now screened at a corrected age of 2 years after birth.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-04; Study Completion 2012-12

CONTACTS AND LOCATIONS:
Overall Officials: Mario Ruediger, Principal Investigator — Technische Universität Dresden
Locations (1):
- University Hospital Carl Gustav Carus, Dresden, Dresden, Germany